CLINICAL TRIAL: NCT06372340
Title: The Development and Application of an Intelligent Diagnosis and Treatment System for Pelvic Floor Dysfunction in Elderly Women
Brief Title: Intelligent Diagnosis and Treatment System for Pelvic Floor Dysfunction in Elderly Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023BJYYEC-217-01
Record Dates: First submitted 2024-04-10; First posted 2024-04-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-01

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence; Diagnosis
Keywords: Urinary incontinence; Pelvic floor muscle; Intelligent diagnosis and treatment system; Elderly female; Pelvic floor dysfunction
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence; Disease

STUDY DESIGN:
Intervention Model Description: The participants will be allocated to experimental group(EG) or the control group(CG). Subjects in the experimental group (EG) will receive personalized pelvic floor muscle training guidance provided by the system, whereas subjects in the control group(CG) will exercise according to the handbook or oral guidance.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessments regarding pelvic floor muscle strength will be conducted by an assessor blind to treatment allocation. The assessor will go through a profound assessment training program. Due to the nature of the intervention neither participants nor care providers can be blinded to allocation, but are strongly inculcated not to disclose the allocation status of the participant at the follow up assessments. An employee outside the research team will feed data into the computer in separate datasets so that the researchers can analyse data without having access to information about the allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised and individualized pelvic floor muscle training (Experimental): Subjects in the experimental group (EG) will accept individualized pelvic floor muscle training under the introduction of skilled clinicians.
  Interventions: Procedure: Personalized pelvic floor rehabilitation program generated by the intelligent diagnosis and treatment system.
- Standard training program (Active Comparator): Subjects in the control group(CG) will accept pelvic floor muscle training according to the handbook or oral guidance
  Interventions: Procedure: Standard pelvic floor muscle training(PFMT) program

INTERVENTIONS:
Procedure: Personalized pelvic floor rehabilitation program generated by the intelligent diagnosis and treatment system. — Utilizing machine learning to process and analyze vast amounts of previously collected data, the investigators will establish an intelligent system that can generate personalized pelvic floor exercise prescription by matching factors such as general clinical information and pelvic floor muscle strength data. The experimental group will receive tailored program, including pelvic floor muscle training with diverse intensity and frequency, electrical stimulation, magnetic stimulation, biofeedback and other treatments. The results will ultimately be compared with those taking standardized pelvic floor muscle training only.
  Arms: Supervised and individualized pelvic floor muscle training
Procedure: Standard pelvic floor muscle training(PFMT) program — Participants will be given handbooks with detailed training program: the basic regimen consists of 3 sets of 8 to 12 contractions sustained for 8 to 10 sec each, performed 3 times a day. Patients should try to do this every day and continue for at least 15 to 20 weeks.
  Arms: Standard training program

SUMMARY:
The aim of this study is to propose an intelligent diagnosis and treatment system for for pelvic floor dysfunction in elderly women. The main question it aims to answer: 1) How can the investigators find out early if older women have different pelvic floor muscle functions? 2）How can the investigators give personalized treatment plans based on differences in pelvic floor function? Participants will be assigned different training programs by the system. The investigators will compare the treatment effects and costs of older women with pelvic floor dysfunction using and not using the system. All the participants will be offered examinations for pelvic floor function and different treatments. All examinations and treatments are non-invasive.

ELIGIBILITY:
Inclusion Criteria:

- Women over 60 years old.

Exclusion Criteria:

* Severe pelvic organ prolapse (POP-Q stage>III)
* History of pelvic floor surgery
* Malignant tumor in pelvic
* Allergic to nickel
* Acute inflammation of pelvic or genital tract
* Subjects who has cognitive impairment and cannot sign an informed consent

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Oxford Scale (MOS) | Baseline, Month 3, Month 6, Month 12
  The modified Oxford scale(Mos) is presently the gold standard used to assess pelvic floor muscle strength. Digital assessment of pelvic floor muscle contraction will be performed by the examiner inserting the index and middle fingers approximately 4 cm into the vagina (only the index finger in the case of very narrow hiatus) and palpating the puborectalis muscle at each side of the vagina during contraction. The Modified Oxford Scale (MOS) was used to rate pelvic floor muscle contraction on a scale of 0-5: 0 = no contraction; 1 = minor muscle 'flicker'; 2 = weak muscle contraction; 3 = moderate muscle contraction; 4 = good muscle contraction and 5 = strong muscle contraction.
Surface Electromyography Data | Baseline, Month 3, Month 6, Month 12
  Pelvic floor muscle(PFM) surface electromyography (EMG) testing is one method for assessing the quantity and quality of PFM function. The electromyograms regarding the contraction and relaxation capacity of the PFM will be recorded simultaneously from electrode probes on perineum and adjacent muscles.

SECONDARY OUTCOMES:
The score of Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | Baseline, Month 3, Month 6, Month 12
  The Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in research and clinical practice across the world. It is used to screen for incontinence, to obtain a brief yet comprehensive summary of the level, impact and perceived cause of symptoms of incontinence. The ICIQ-UI SF score ranges from 0 to 21. A score of zero means no leakage of urine and no affection on quality of life.
The score of the Pelvic Floor Distress Inventory (PFDI-20) | Baseline, Month 3, Month 6, Month 12
  The Pelvic Floor Distress Inventory (PFDI-20) is a patient-reported outcome measures that is often used in clinical practice and clinical trials to assess the distress caused by the presence of pelvic floor dysfunction. It assesses the distress of pelvic organ prolapse (POP), anorectal and urinary symptoms in three subscales, respectively. PFDI-20 summary score ranges from 0 to 300. It is interpreted as the higher the score, the worse the distress.
Subjective staging used Pelvic Organ Prolapse Quantification (POP-Q) System | Baseline, Month 3, Month 6, Month 12
  The POP-Q describes descent of the anterior and posterior vaginal wall and uterine cervix or, after hysterectomy, the vaginal vault, relative to the hymen on maximal Valsalva maneuver. In clinical practice, the POP-Q is often used to stratify findings into stages - Stage 0 (normal) and Stages 1-4 (prolapse).

CONTACTS AND LOCATIONS:
Overall Officials: Mi Li, Ph.D., Study Chair — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in pelvic floor muscle dysfunction. Data or samples shared will be coded, with no protected health information (PHI) included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial individual participant data (IPD) can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact mindy99999@126.com.